CLINICAL TRIAL: NCT06481878
Title: Validation of a Diagnostic and/or Prognostic Marker for Alzheimer's Disease by Fecal Determination of Amyloid Peptides and Tau Proteins
Brief Title: Validation of an Alzheimer's Disease Marker by Fecal Assay of Amyloid Peptides and Tau Proteins
Acronym: FecAlz
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC24.0026; 2024-A00378-39 (Other: ID RCB)
Record Dates: First submitted 2024-05-31; First posted 2024-07-01 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Occult Blood

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Feces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 35 MA TCM (A+ T+): Group of patients with established Alzheimer's disease at the stage of major cognitive impairment
  Interventions: Diagnostic Test: faecal analysis
- 15 MA TCm (A+ T+): Group of patients with established Alzheimer's disease at the stage of minor cognitive impairment
  Interventions: Diagnostic Test: faecal analysis
- 15 TC Non MA LCR negatif (A- T-): Group of patients with minor or major cognitive impairment but without AD
  Interventions: Diagnostic Test: faecal analysis
- 15 TCm LCRdiscordant (A+ T-) ou (A- T+): Group of patients with minor cognitive impairment and discordant CSF
  Interventions: Diagnostic Test: faecal analysis
- 35 VS: Group of healthy volunteers
  Interventions: Diagnostic Test: faecal analysis

INTERVENTIONS:
Diagnostic Test: faecal analysis — Collection of medical data and stool sampling

SUMMARY:
Alzheimer's disease (AD) is the leading cause of dementia in humans, currently affecting almost one million people in France. It results from an irreversible degeneration of neurons responsible for a progressive decline in the main cognitive and memory functions due to a cerebral accumulation of plaques containing fibrillary amyloid peptide (Aβ) and neurofibrillary tangles composed of truncated, hyperphosphorylated tau protein (pTau).

There is currently no curative treatment for this disease in France. However, two treatments aimed at reducing beta-amyloid plaques in the brain have been approved by the U.S. Food and Drug Administration. The failure of the latest therapeutic strategies is largely due to the fact that the disease is diagnosed too late, starting with a long asymptomatic phase, which is the one that needs to be targeted in order to prevent irreversible neurodegenerative mechanisms.

The development of diagnostic tools is gradually making it possible to detect such a sequence, but this has its drawbacks (radioactive load, invasive procedure, cumbersome set-up).

Over the last ten years, research has focused on the development of plasma or salivary markers. Although encouraging, these studies show either a lack of sensitivity or reproducibility, or a lack of specificity or precocity.

The expression of Aβ and Tau proteins has recently been demonstrated in the enteric nervous system and enterocytes. Intestinal Aβ is involved in various gut functions and regulation.

What recent work by investigators demonstrates is the essential and hitherto unrecognized role of the gut-brain axis in maintaining brain homeostasis. In a mouse model of AD, the investigators have demonstrated a mechanism for intestinal elimination (clearance) of toxic brain forms of Tau and Aβ proteins, via the lymphatic network.

The clearance of cerebral Tau and Aβ proteins in the stool may constitute a reliable and powerful diagnostic signature of AD. Its study would represent a new, non-invasive and easily accessible technique for the early diagnosis of AD in humans.

ELIGIBILITY:
Inclusion Criteria:

For subjects with Alzheimer's disease MA TCM (A+ T+):

* Subjects diagnosed with AD according to IWG 2021 criteria
* Subject at the stage of major cognitive impairment
* At least 40 years of age
* Presence of a caregiver or support person
* No informed opposition

For subjects with AD TCm (A+ T+):

* Subject diagnosed with AD according to IWG 2021 criteria
* Subject at the stage of minor cognitive impairment
* Minimum age 40
* No informed opposition For subjects with minor or major cognitive impairment who do not have AD TC Non-AD LCR negative (A- T-)
* Subject at stage of minor or major cognitive impairment
* CSF negative (A-T-) for Alzheimer's disease biomarkers: A-T- according to ATN classification
* Minimum age 40
* No informed objection and TCm CSFdiscordant (A+ T-) or (A- T+):
* Subject at stage of minor cognitive impairment
* CSF discordant (A-T+ or A+T-) with Alzheimer's disease biomarkers
* Minimum age 40
* No informed opposition

For healthy volunteers (VS) :

* No cognitive complaints
* MMSE ≥ 26
* CDR 0
* Minimum age 40
* No informed opposition

Exclusion Criteria:

For MA TCM (A+ T+), MA TCm (A+T+) and TC Non MA LCR negatif (A-T-) and TCm LCRdiscordant (A+ T-) or (A- T+):

* Inability to understand search instructions or to give informed non-opposition
* Absence of social security affiliation or plan
* Persons covered by articles L1121-5 to L1121-8 of the CSP (legally protected adult, subject under administrative or judicial supervision)

For healthy volunteers:

* Incapacity to understand research instructions or to give informed non-opposition
* Persons covered by articles L1121-5 to L1121-8 of the CSP (legally protected adult, subject under administrative or judicial supervision)
* Absence of social security affiliation or of such a scheme

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Single-center study, recruitment among patients consulting the CMRR of the Alpine arc
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2027-10-06 (Estimated); Study Completion 2027-10-06 (Estimated)

PRIMARY OUTCOMES:
to determine the amount of fibrillar and oligomeric amyloid peptide and phosphorylated tau protein measured in the stools of subjects issued as soon as possible after recruitment | Between inclusion and Month 6
  Quantity of AD biomarkers in stool.
  The biomarkers studied will be :
  In Lumipulse (CHUGA platform): beta-amyloid 42,beta-amyloid 40, Ptau and total tau.
  Dotblot (GIN): Soluble forms of phosphorylated tau (Tau-pThre205, Tau-pThre181, Tau-pThre217, Tau-pser404) or total tau (panTau), as well as toxic oligomeric forms of the beta-amyloid peptide (E22P). Finally, insoluble fibrillar forms of Tau (AT8) and beta-amyloid peptide (OC).

SECONDARY OUTCOMES:
To observe the evolution and kinetics of AD biomarkers in subjects with Alzheimer's disease at the stage of minor cognitive impairment (AD TCm A+ T+). | between Month 6 and Month 12
  Quantity of AD biomarkers in the stool of subjects with Alzheimer's disease at the TCm stage between M6 and M12 (AD TCm A+ T+)
Follow the efficacy of a treatment if the AD TCm (A+ T+) subject takes one | between Month 6 and Month 12
  Increase or decrease in the quantity of AD biomarkers in the stool of subjects with Alzheimer's disease at the TCm stage under treatment between M6 and M12 (AD TCm A+ T+).
Observe the evolution and kinetics of AD biomarkers in subjects without Alzheimer's disease at the stage of minor cognitive impairment (TCm LCRdiscordant). | between Month 6 and Month 12
  Quantity of AD biomarkers in the stool of non-Alzheimer's subjects at stage TCm CSFdiscordant) between M6 and M12

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde SAUVEE, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Grenoble Alpes University Hospital, Grenoble, France